CLINICAL TRIAL: NCT05326126
Title: Microvascular Function in Patients Undergoing Transcatheter Aortic Valve Implant (TAVI) for Severe Symptomatic Aortic Stenosis: Association With Myocardial Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matteo Montorfano (Other)
Responsible Party: Sponsor-Investigator, Matteo Montorfano, Interventional cardiologist, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAVI IMR
Record Dates: First submitted 2021-10-08; First posted 2022-04-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Severe Symptomatic Aortic Stenosis

STUDY DESIGN:
Intervention Model Description: TAVI's intervention will be performed as per current clinical indications and according to the hospital's clinical practice. To this will be added the evaluation of coronary physiology using Pressure Eire X and Coroventis software, which, although performed in accordance with the IFU of the aforementioned devices, is considered an experimental procedure. Adenosine will be required to complete the measurement of coronary physiology
Masking Description: Patients will be assigned a univocal identification code. Medical personnel in charge of baseline, in-hospital and follow-up data acquisition will be allowed to know each patient identity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Coronary physiology evaluation (Experimental): Patient will undergo TAVI and then Myocardial fibrosis will be evaluated on images acquired at the time of the cardiac CT obtained for TAVI planning. Briefly, an extra late post-contrast acquisition image will be acquired. The delayed post-contrast scan will be reconstructed with a soft convolution kernel and will be reformatted in the short- and long-axis planes (slice thickness 8 mm; gap 0 mm) in average mode.
  Interventions: Device: coronary physiology

INTERVENTIONS:
Device: coronary physiology — To evaluate the association between microvascular disfunction and myocardial fibrosis identified per computed tomography among subjects undergoing TAVI for severe, symptomatic aortic stenosis.

SUMMARY:
Microvascular function in patients undergoing Transcatheter Aortic Valve Implant (TAVI) for severe symptomatic aortic stenosis: association with myocardial fibrosis

DETAILED DESCRIPTION:
Severe symptomatic aortic stenosis is commonly encountered in clinical practice, affecting close to 5% of individuals older than 65 years of age, and carries a dismal prognosis if left untreated.(1,2) Chronically increased left ventricular afterload triggers a compensatory myocardial response, ultimately leading to ventricular hypertrophy, aimed at reducing chronically increased wall tension an restore cardiac performance.(3) Hypertrophy ultimately results in maladaptive changes and ultimately leads to heart failure and eventually increased risk of cardiac mortality. Myocardial fibrosis and altered myocardial perfusion appear to play a role in progressive cardiac decompensation.

ELIGIBILITY:
Inclusion Criteria:

• All patients referred to IRCCS Ospedale San Raffaele who are candidates to receive a TAVI implant for severe, symptomatic aortic stenosis under current appropriateness criteria and clinical practice guidelines will be considered eligible to take part in the study

Exclusion Criteria:

* Age <18 years
* Inability to express informed consent to take part in the present study.
* Pregnancy or lactation
* Pre-existing known disease determining a prognosis quo ad vitam shorter than the follow up of the present study
* Significant chronic kidney disease (estimated glomerular filtration rate <30 ml/min)
* Known significant epicardial coronary artery stenosis
* Known contraindication to adenosine administration:
* Known allergic reactions
* Second or third degree atrioventricular block before the procedure (in absence of a functional permanent pacemaker)
* Long QT syndrome
* Unstable angina
* Severe hypotension
* Acutely decompensated heart failure
* Chronic obstructive pulmonary disease with bronchospasm
* Concomitant use of dypiridamole

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
The burden of myocardial fibrosis | 1 year
  Myocardial fibrosis measured as the percentage of delay-enhanced myocardium over total myocardial volume
Index of microcirculatory resistance (IMR) | 1 year
  IMR a validated estimate of resistance in the coronary capillary, computed as the ratio between transit time of a 3 cc bolus of room temperature saline and distal coronary artery pressure.

SECONDARY OUTCOMES:
Acute change in coronary flow reserve (CRF) | 1 year
  Ratio of maximal coronary blood flow obtained by hyperemia to baseline coronary blood flow
Acute change in index of microcirculatory resistance (IMR) | 1 year
  Estimate of microvascular resistance derived by pressure and an indirect estimate of flow
Computed tomography derived extracellular volume | 1 year
  The extracellular volume fraction (ECV) is the relative value of the volume of the extracellular space in the myocardium, therefore express as a percentage. It could be measured from computed tomography (CT) and Index of microcirculatory resistance (MRI) images, and was validated with histology. ECV-CT is calculated as follows:
  ECVCT = (1-haematocrit) × (ΔHUmyo/ΔHUblood) where ΔHU is the change in Hounsfield unit attenuation pre- and post-contrast (i.e. HUpost-contrast - HUpre-contrast)
All-cause death | 1 year
  Death from any cause
Cardiovascular death | 1 year
  Death from any cardiac condition (e.g. myocardial infarction, acute pulmonary edema, low-output state, etc..) or vascular condition (including aortic dissection, stroke, etc…)
Any rehospitalization | 1 year
  Admission to an inpatients' service for any cause lasting >24h
Cardiovascular rehospitalization | 1 year
  Admission to an inpatients' service for cardiovascular conditions lasting >24h

CONTACTS AND LOCATIONS:
Overall Officials: Matteo montorfano, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No